| Official Title: | Moving PD-1 Blockade with Pembrolizumab into |
|---|---|
| | Concurrent Chemoradiation for Locally Advanced Non- |
| | Small Cell Lung Cancer (Multi-Center) |
| NCT number: | 02621398 |
| <b>Document Type:</b> | Study Consent - Main |
| Date of the | 08/29/2 <b>018</b> |
| Document: | |



This consent form is part of an informed consent process for a research study and it will provide information that will help you to decide whether you wish to volunteer for this research study. It will help you to understand what the study is about and what will happen in the course of the study.

If you have questions at any time during the research study, you should feel free to ask them and should expect to be given answers that you completely understand.

The study doctor,
given a copy of the signed consent form to keep.

You are not giving up any of your legal rights by volunteering for this research study or by signing this consent form.

Even after signing this consent form, you may withdraw from the study at any time.

Sponsor of the study

supply the study drug, is the sponsor of this study.

and is providing funding support.

#### Why is this study being done?

This study is being done to test the good and bad effects of the study drug called pembrolizumab when given during and/or after completion of your chemotherapy and radiation. Giving you this medication after or in combination with chemotherapy and radiation may increase the amount of time your disease is not active or does not spread to another part of your body.

Pembrolizumab is a PD-1 inhibiting drug and has been approved by the FDA to treat melanoma and other medications in this class of PD-1 drugs have been also approved for lung cancer. Typically, the human body's immune system recognizes abnormal cells in the body and destroys them. Cancer cells frequently create proteins on the cell surface (PD-L1) that act as signals to turn off this part of the immune system. Pembrolizumab is a drug that blocks (inhibits) this signal on the immune system's cells (PD-1) and allows the immune system to recognize these cancer cells as foreign.

in this study is investigational. "Investigational" means that this medication has not yet been approved by the FDA to treat the type of cancer you have. Your voluntary participation in this research study may help to find out whether the PD-1 inhibiting drug, pembrolizumab, is effective at lengthening the time until your cancer starts to grow.

The purpose of this study is to:

- 1) To determine the good and bad effects of adding pembrolizumab after completing or while receiving chemotherapy and radiation;
- To determine what dose of pembrolizumab is safe to give in combination with chemotherapy and radiation. Dose escalation determines the least toxic and most effect dose of this drug combination for treatment.

#### Why have you been asked to take part in this study?

You are being asked to take part in this study because you have inoperable non-small cell lung cancer (NSCLC). People who complete their treatment are usually observed on a regular basis for progression of their disease.

### Who may take part in this study? And who may not?

You may take part in this study if you are 18 years of age or greater with inoperable non-small cell lung cancer. Additionally, you may take part in this study if:

- Your treatment plan includes chemotherapy and radiation
- You have tumor available from a recent surgery or biopsy
- · You have read and signed this Informed Consent Form

You may not take part in this study if:

- You have cancer that has spread outside the lungs to other parts of the body
- · You are unable to keep your doctor's appointments
- You are pregnant or breast feeding

## How long will the study take and how many subjects will participate?

You will receive chemotherapy and radiation therapy for 6 weeks. Study treatment with pembrolizumab will continue for one year, as long as your tumor is responding and you are not experiencing severe side effects. After you have stopped receiving treatment on study, we will continue to follow up with you for the rest of your life.

A total of approximately 30 patients will take part in this study. You will be one of approximately 10 patients enrolled at the

## What will you be asked to do if you take part in this research study?

Before you begin study treatment:

You will have some exams, tests and procedures to find out if you can take part in this study. Most of the exams, tests, and procedures you will have are part of the usual approach for your cancer. However, your doctor will do some extra testing as part of the study. The testing that you will need to have if you take part in this study is discussed below. If some of these have been done recently they may not need to be repeated, this will be up to the study doctor.

- Your age and race/ethnicity will be recorded.
- You will be asked about your medical history and any medications you are currently taking, both prescription and over the counter.

- a complete physical examination, with your physician or physician's assistant, including measurement of your vital signs (breathing rate, blood pressure, temperature, and heart rate), height, and weight.
- Evaluation of your ability to carry out daily activities.
- The following blood samples will be collected within 14 days of registration:
  - Approximately 2 teaspoons (10 mL) for routine testing, such as, a complete blood count, kidney and liver function tests to ensure that it is safe to administer any of the drugs included in this study
  - Approximately 1 teaspoon (5 mL) for blood clotting tests
  - o Approximately 1 teaspoon (5 mL) for thyroid function testing
- If you are a woman who could become pregnant (even if you had a tubal ligation), your
  doctor will perform a blood or urine pregnancy test. If you are pregnant, you cannot
  participate in this study.
- · Pulmonary Function Tests, to see how well the lungs work
- Imaging tests typically performed for cancer patients, including imaging of chest, abdomen and brain. Scans will include:
  - Computed tomography (CT), a scan that uses x-rays to look at one part of your body. It may be done with or without contrast. Contrast means that dye is injected into your vein to increase the differences between normal and abnormal tissue.
  - Magnetic resonance imaging (MRI), imaging that uses a strong magnetic field to look at one part of your body.
  - Operation Positron emission tomogram (PET), uses computerized images to look at the activity of tumor cells in your entire body and that requires injection of a special marker into your vein, such as sugar (glucose) combined with a low-dose radioactive substance (a tracer). A camera records the tracer's signal as it travel through your body.
- You will be asked to provide a sample of your tumor for research from a recent surgery
  or biopsy (within 8 weeks). If your tumor specimen is greater than 8 weeks old, you may
  still be able to take part in the study if the tumor is available, the sponsor gives
  permission and you are willing to undergo a fine needle aspiration (a method to remove a
  piece of lung tissue for examination).

Your doctor will send the tumor sample to a central lab for testing of certain proteins and biomarkers (indicators of normal biological or disease processes) that may be involved in PD-1 activation or to understand the nature of your disease. These laboratory tests are new and under development. Any remaining slides after the testing is completed will be destroyed.

If you do not meet the eligibility requirements, you cannot take part in this study. The study doctor will inform you of other options that are available to you.

#### STUDY TREATMENT

If the tests, exams, procedures show that you can be in the study, you will be registered. All study participants will receive chemotherapy (paclitaxel and carboplatin), radiation therapy and pembrolizumab.

- <u>Radiation Therapy:</u> You will receive radiation therapy daily (Monday Friday) for 6 weeks. Each treatment may take up to 15-30 minutes depending on the technique used.
- <u>Chemotherapy</u>: You will start chemotherapy the same day as you start radiation therapy
  and then receive chemotherapy once a week. You will receive chemotherapy before your
  radiation treatment on days you are scheduled to receive both.
- <u>Pembrolizumab</u>: Depending on what part of the study you enter, the dose and time when you start treatment with pembrolizumab will vary. The timing of this medicine could be after or during the radiation therapy.

### Radiation Therapy:

Your study doctor will decide what type of radiation therapy you will receive.

- 3-Dimensional conformal radiation therapy or intensity modulated radiation therapy (IMRT) is a form of radiation in which a number of x-ray beams are used to shape the radiation to the cancer and is designed to avoid important normal parts of your body.
- Image guided radiation therapy (IGRT) radiation part of the routine radiation treatment that
  helps to align the radiation accurately to the tumor. Small adjustments in your radiation
  treatment are made each treatment day based on x-ray images taken right before each day's
  treatment to ensure that your radiation treatment is given as accurately as possible.
- Proton Beam Therapy (PBT) is another type of external radiation treatment and is precise like IMRT, but uses proton beams instead of x-ray beams to direct the radiation.

Before you begin radiation therapy, you will have imaging of the chest in order to design your radiation treatment. Doctors will use information gathered from these scans to plan the best way to deliver radiation to your tumor.

#### Chemotherapy:

You will receive paclitaxel and carboplatin once a week starting with radiation therapy. On days you are scheduled to receive both, you will receive chemotherapy prior to radiation therapy. Paclitaxel will be given intravenously (IV) through a vein over 1 hour; followed by carboplatin, given IV over 30 minutes. You will receive pre-medication to reduce side effects related to chemotherapy such as nausea and vomiting.

#### Pembrolizumab:

The dose and time of when you start treatment with pembrolizumab will vary based on when you enter the study. Below is a table of the different parts of the study. Pembrolizumab will be given Day 1 of every 3 week cycle. It will be given by IV through a vein over 30 minutes. Treatment with pembrolizumab will continue for up to 12 months for as long your disease is not growing and you are tolerating treatment.

| Part | Start of Pembrolizumab | Dose of Pembrolizumab |
|---|---|---|
| 1 | 2-6 weeks after completing chemotherapy and radiation | 200 mg |
| 2 | Week 5 of chemotherapy and radiation | 100 mg |
| 3 | Week 5 of chemotherapy and radiation | 200 mg |
| 4 | Week 1 of chemotherapy and radiation | 100 mg |
| 5 | Week 1 of chemotherapy and radiation | |

## While on study treatment:

During the treatment period, you will need the following examinations, tests, and procedures described below. Some of these exams, tests, and procedures are part of your regular medical care.

You will have the following done weekly while receiving chemotherapy and radiation therapy, then on Day 1 of every 21 day cycle while receiving pembrolizumab alone:

- You will be asked to report any symptoms and health problems you have and any new medications you have started.
- You will have a complete physical examination, with your physician or physician's
  assistant, including measurement of your vital signs (breathing rate, blood pressure,
  temperature, and heart rate), height, and weight.
- Evaluation of your ability to carry out daily activities.
- · You will have blood tests:
  - Approximately 2 teaspoons (10 mL) for routine testing, such as, a complete blood count, kidney, and liver function tests.
  - Approximately 1 teaspoon (5 ml) for thyroid function tests every 3 weeks while receiving pembrolizumab
- On days 8 and 15 of every 21 cycle of Pembrolizumab you will be asked to report any symptoms and health problems you have and any new medications you have started, this may be done by a phone call.
- Tumor Assessments: You will have a CT scan of the chest and/or abdomen every 9 weeks while receiving pembrolizumab to evaluate how your cancer is responding to the cancer.
- Research Labs: In addition to blood tests required to monitor your health, other blood
  tests will be done to see how the immune system responds to the different treatment
  combinations and doses. An additional 2 teaspoons (10 mL) will be collected during
  weeks 1, 3, and 6 of chemotherapy and radiation and during Cycle 1, 2 and 3 of
  pembrolizumab. These labs are being done for study only. They will be sent to a central
  laboratory for testing and will not be a part of your medical record.

## After you have completed study treatment:

Your doctor will stop study treatment if any of the following occur:

- Your tumor grows larger or you develop new tumors (disease progression)
- You develop unacceptable side effects
- You become pregnant or are unwilling to use appropriate birth control techniques
- The study doctor determines that it is not in your best interest to continue the study treatment
- You have completed study treatment as planned and your disease has not worsened
- · New information becomes available
- The study is stopped by the

& the IRB or FDA

You choose to stop study treatment

After all study treatment has stopped, your doctor will ask you to return to the clinic for an end of treatment visit, which will be approximately 30 days after your last dose of study drug. You will return for another clinic visit approximately 8 weeks after your last dose of study drug. The following assessments will be done at these visits:

- You will be asked to report any symptoms and health problems you have and any new medications you have started.
- You will have a complete physical examination, with your physician or physician's
  assistant, including measurement of your vital signs (breathing rate, blood pressure,
  temperature, and heart rate), height, and weight.
- Evaluation of your ability to carry out daily activities.
- If you have any remaining side effects after treatment, you may have blood tests (at the 30 day post-treatment visit):
  - Approximately 2 teaspoons (10 mL) for routine testing, such as, a complete blood count, kidney, and liver function tests.

#### Follow-Up

If you have any ongoing side effect at the time you complete the study or your doctor discontinues you from the study, the study doctor will continue to follow your condition until the side effect resolves or becomes stable.

You will have imaging tests every 12 weeks for the first year, then every 16 weeks for the second year and then every 6 months for years 3-5.

If your disease worsens or you withdraw from the study treatment but not from study follow-up, the study staff will contact you approximately every 12 weeks after your last visit to check on your health status. If they are not able to reach you, they may use a public information source (like county records) to obtain information about your survival status only, which will be reported as part of the data for the study.

#### **Second Course Treatment:**

You may be eligible for up to one year of additional pembrolizumab (MK-3475) therapy if the disease progresses after stopping pembrolizumab (MK-3475). Your study doctor will determine if you meet the study criteria to be eligible for the Second Course Treatment. If you are eligible, you will restart treatment at the dose and dose frequency received upon initial treatment with pembrolizumab (MK-3475).

What are the risks and/or discomforts you might experience if you take part in this study? You may have side effects from the drugs or procedures used in this study, and they will vary from person to person. Study doctors will carefully watch everyone taking part in the study for any side effects. However, the study doctors and the study funders do not know all the side effects that may happen, and unknown side effects that could occur. The study doctors may give you medicine to help lessen the side effects. In some cases, side effects can be serious, long lasting, and/or may never go away. There also is a rare risk of death. You should talk to your study doctor about any side effects that you have while taking part in the study.

If you experience any severe side effect, you should:

• Seek professional medical help immediately



- Call your study doctor
- · If necessary, go to the nearest emergency room

#### Possible Side Effects of Paclitaxel

Common, Some may be Serious (in 100 people receiving Paclitaxel, more than 20 and up to 100 may have):

- · Anemia which may cause tiredness, or may require blood transfusions
- · Infection, especially when white blood cell count is low
- Diarrhea, nausea, vomiting
- Sores in mouth which may cause difficulty swallowing
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Bruising, bleeding
- Pain
- Muscle weakness
- Numbness, tingling or pain of the arms and legs
- Hair loss

# Occasional, Some may be Serious (in 100 people receiving Paclitaxel, from 4 to 20 may have):

- Abnormal heartbeat
- Damage to the lungs which may cause shortness of breath
- · Blood clot which may cause swelling, pain, shortness of breath

#### Rare, and Serious (in 100 people receiving Paclitaxel, 3 or fewer may have):

- Heart attack or heart failure which may cause shortness of breath, swelling of ankles, and tiredness
- A tear or a hole in the stomach which may cause belly pain or that may require surgery

#### Possible Side Effects of Carboplatin

Common, Some may be Serious (in 100 people receiving Carboplatin, more than 20 and up to 100 may have):

- Hair loss
- Vomiting, nausea
- Infection, especially when white blood cell count is low
- Anemia which may cause tiredness, or may require blood transfusions
- Bruising, bleeding
- Belly pain

# Occasional, Some may be Serious (in 100 people receiving Carboplatin, from 4 to 20 may have):

- · Diarrhea, constipation
- Numbness and tingling in fingers and toes



 Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat

### Rare, and Serious (in 100 people receiving Carboplatin, 3 or fewer may have):

- Changes in vision
- Changes in taste
- Damage to organs which may cause hearing and balance problems

#### Possible Side Effects of Lung Radiation

Common, Some may be Serious (in 100 people receiving lung radiation treatment, more than 20 and up to 100 may have):

- Swelling and redness, tanning, thickening, numbness, or peeling of the skin in the area of radiation
- Difficulty and/or pain with swallowing
- Hair loss in the treatment area, may be permanent
- · Shortness of breath
- Cough with or without increased phlegm production
- Tiredness
- Diarrhea, nausea

# Common, Some may be Serious (in 100 people receiving lung radiation treatment, more than 20 and up to 100 may have):

- · Anemia, which may require blood transfusion
- Infection, especially when white blood cell count is low
- Bleeding, bruising
- Rib pain, increased risk of rib fracture

# Occasional, Some may be Serious (in 100 people receiving radiation treatment, from 4 to 20 may have):

- Inflammation of the lung that may cause difficulty breathing and can be life-threatening
- Narrowing of the throat which may cause vomiting, difficulty swallowing
- Scarring in the lung
- Lung collapse
- Fluid around lungs
- Bleeding from the lungs which may cause coughing up blood
- Fever
- Narrowing of the esophagus
- Pain in chest wall

#### Side Effects of Pembrolizumab

Pembrolizumab which is approved in the *USA and* some other countries is available by prescription to treat several different cancers, but may not be approved to treat your type of cancer.



Overall, as of 03-Mar-2018, approximately 25,519 patients have been treated with pembrolizumab in clinical studies.

Pembrolizumab works by helping your immune system to fight your cancer.

However, pembrolizumab can also cause your immune system to attack normal organs and tissues in your body and can affect the way they work, which can result in side effects. These side effects may be serious (i.e., causing hospitalization or be life threatening) and may result in death, and/or may occur after you stop taking pembrolizumab.

#### Very Common

Out of 100 people who receive pembrolizumab, 20 or more people may have the following:

- Itching of the skin
- · Loose or watery stools
- Cough

#### Common

Out of 100 people who receive pembrolizumab, at least 5 but less than 20 people may have the following:

- Joint pain
- Fever
- Back pain
- Rash
- Pain in your belly
- Loss of skin color
- Not enough thyroid hormone so you may feel tired, gain weight, feel cold, have infrequent or hard stoolsLow level of salt in the blood that may cause you to feel tired, confused, have a headache, muscle cramps and/or feel sick to your stomach

#### Uncommon

Out of 100 people who receive pembrolizumab, at least 1 but less than 5 people may have the following:

- Inflammation of the lungs; so you may feel short of breath and cough.
- Too much thyroid hormone so you may feel anxious, angry, have trouble sleeping, feel weak, tremble, sweat, feel tired, have loose and watery stools
- Infusion reaction, where you may feel dizzy or faint, flushed, get a rash, have a fever, feel short of breath at the time of receiving your infusion (IV) or just after, or pain at the site of infusion
- Inflammation of the bowels/gut, which may cause severe pain in your belly with loose or watery stools and black, tarry, sticky stools or stools with blood or mucus



Inflammation of the skin so you may have peeling of the skin, itchiness and/or skin
redness. The skin inflammation (i.e. peeling, itching, and redness) could also be
widespread throughout your body. More severe skin reactions may involve the inside of
your mouth, the surface of your eye and genital areas, and/or may cause the top layer of
your skin to peel from all over your body which can cause severe infection.

#### Rare

# Out of 100 people who receive pembrolizumab, less than 1 person may have the following:

- Inflammation of the nerves that may cause pain, weakness or tingling your hands and feet, and may spread to your legs, arms and upper body leading to severe muscle weakness and possible temporary paralysis.
- Inflammation of the muscles so you may feel weak or have pain in your muscles
- Inflammation of the pancreas (a gland in your abdomen that controls sugar levels) so you
  may have severe upper abdominal pain that may move to your back, feel sick to your
  stomach, and vomiting that gets worse when you eat
- Inflammation of the eye so you may have eye redness blurred vision, sensitivity to light, have eye pain, see floaters or have headaches
- Inflammation of the liver that may make you feel sick to your stomach and vomit, feel like not eating, feel tired, have a mild fever, have a pain in the right side your belly, yellow eyes and skin, and dark urine
- Inflammation of the pituitary gland (a gland in the head), which may cause you to feel
  sick to your stomach or have headaches changes in your behavior, double vision, few to
  no menstrual cycles, weakness, vomiting and dizziness or fainting.
- Adrenal glands (glands on top of the kidneys) that may not make enough hormone which
  could cause tiredness, weight loss, muscle weakness, feeling faint, joint, muscle and belly
  aches, nausea, vomiting, diarrhea, fever, salt craving, and sometimes darkening of the
  skin like a suntan.
- Type 1 Diabetes, a condition that can cause too much sugar in your blood, feeling thirstier than usual, frequent urination and weight loss. You are likely to need regular insulin shots.
- Inflammation of the kidney so you may pass less urine or have cloudy or bloody urine, swelling and low back pain
- Too much sugar in your blood (diabetes), so you may feel thirsty, and may need regular
  insulin shots.
- Inflammation of the middle layer of your heart wall that may cause your heart to have difficulty pumping blood throughout your body, which can cause chest pain, shortness of breath and swelling of the legs. You may experience a fast or irregular heartbeat that may cause dizziness or fainting. Inflammation of the thyroid gland, an organ that makes and stores thyroid hormones. This condition may lead to change in your heart rate, blood pressure, body temperature, and the rate at which food is converted into energy.
- A condition that may make you feel weak and tired and might have drooping of the
  eyelids, blurred or double vision, difficulty swallowing, slurred speech, weakness in your
  arms and legs, or difficulty breathing.
- The formation of small clusters of immune cells (called granulomas) in parts of your body such as your lymph nodes, eyes, skin, or lungs

the brain with confusion and fever. This may also include: disorientation, memory problems, seizures (fits), changes in personality and behavior, difficulty speaking, weakness or loss of movement in some parts of your body, and loss of consciousness

Additionally, since pembrolizumab was approved in September 2014, the following side effects have been reported by people receiving pembrolizumab. These side effects were voluntarily reported from a group of people of unknown size. It is not possible to estimate the frequency of this side effect:

• Inflammation of the joints which may include joint pain, stiffness and/or swelling

If you have had an allogeneic stem cell transplant (a procedure in which a person receives blood-forming stem cells from a donor), you may experience graft versus host disease (GvHD), which may include diarrhea, skin rashes, and liver damage, after receiving pembrolizumab. Sometimes this condition can lead to death.

If you have had a solid organ transplant (for example, if you have received a kidney or heart transplant), you may experience rejection of the transplanted organ. Your doctor will monitor you and should tell you what signs and symptoms you should report depending on the type of organ transplant that you have had.

Patients treated with pembrolizumab **BEFORE** going on to receive an allogeneic stem cell transplant (a procedure in which a person receives blood-forming stem cells from a donor), should inform their transplant physicians that they have received pembrolizumab in the past.

In patients with any hematologic malignancy (cancers of the blood like Hodgkin lymphoma, multiple myeloma): there is a potential for an increased risk of severe complications following allogeneic stem cell transplant in patients who previously received pembrolizumab **BEFORE** an allogeneic stem cell transplant.

Reports of clotting of blood within the liver and severe graft versus host disease (which can include skin, liver and gastrointestinal symptoms), including death, have been received for patients who received pembrolizumab **BEFORE** an allogeneic stem cell transplant.

Patients with multiple myeloma who were treated with pembrolizumab in combination with either pomalidomide or lenalidomide (drugs related to thalidomide which affect the body's immune system) and dexamethasone (a steroid) had an increased number of serious side effects and deaths as compared to patients who received only dexamethasone and either pomalidomide or lenalidomide.

#### Reproductive risks

You should not become pregnant or father a baby while on this study because the drugs and radiation treatment in this study can affect an unborn baby. Women who are able to have children will have a pregnancy test before beginning treatment. Women should not breastfeed a baby while on this study. It is important you understand that you need to use birth control for as

treatment on this study and for 120 days after completion of all treatment to prevent pregnancy or fathering a child. Check with your study doctor about what kind of birth control methods to use. Some methods might not be approved for use in this study. The treatment in the study may make you unable to have children in the future. Women of childbearing age can ask their doctor for information about pre-treatment or post-treatment reproductive or fertility options prior to agreeing to participate in the study.

#### Possible Risks Related to Reproductive health/sexual activity

Researchers have not studied the effect of the study drug, pembrolizumab, on human sperm and eggs. They also do not know the effects on the developing fetus using the study drug during pregnancy and the risk of birth defects from use of pembrolizumab. Therefore, both men and women should not attempt pregnancy and women should not be pregnant or breast-feeding while taking part in this study and for at least 120 days after your last dose of the study drug pembrolizumab.

If sexually active, both men and women should use an effective method of birth control while taking the study drug. Barrier contraceptives (condoms or diaphragm) with spermicide, intrauterine devices (IUDs), hormonal contraceptives, oral contraceptive pills, surgical sterilization, and complete abstinence are examples of effective methods. Only methods that use condoms provide reasonable/true protection against sexually transmitted diseases. If you or your partner become pregnant while taking the study drug, you must tell your study nurse/doctor immediately. You may have to stop the study drug. Your doctor will discuss other treatment options with you if you stop the study drug.

A woman should not breast-feed a baby while in this study because pembrolizumab may enter the breast milk and possibly harm the child.

If you are a woman capable of bearing children, you will have a pregnancy test before you can participate in this study. If at any time during the study or within 120 days after your last dose of the study drug pembrolizumab you suspect that you have become pregnant, please notify the study doctor immediately.

Male participants should immediately inform the study doctor if your partner becomes pregnant during the study, within 120 days after your last dose of the study drug pembrolizumab.

### Are there any benefits for you if you choose to take part in this research study?

Taking part in this study may or may not make improve your health better or allow you to live longer. The information from this study will help doctors learn more about pembrolizumab as a treatment for NSCLC. This information could help other people who have a similar medical condition in the future.

#### What are your alternatives if you don't want to take part in this study?

You do not have to take part in this research study. If you decide not to take part in this study, you have other choices. Instead of being in this study, you can:

- Choose to have the usual approach to treatment described above without being in a study
- Take part in another study
- Get comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems, and other problems caused by the cancer. It does not treat

the cancer directly, but instead tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.

Please talk to the study doctor about your choices before you decide if you will take part in this study.

# How will you know if new information is learned that may affect whether you are willing to stay in this research study?

During the study, your study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study. When informed of this new information, if you agree to continue in the study, your doctor will ask you to sign an updated Informed Consent Form.

### Will there be any cost to you to take part in this study?

You will have tests and procedures that are part of your regular medical care (not part of the research), including the treatment with chemotherapy and radiation therapy. You or your insurance company or third party provider will be responsible for these costs, including copayments and deductibles.

The study will provide the drug pembrolizumab at no charge to you while you take part in this study. The study does not pay for the cost of getting the study drug ready and giving it to you intravenously (in a vein). You or your insurance company will pay for this procedure.

Your doctor and your other health care providers will bill the cost of your regular medical care to you or to your health insurance company in the usual way. However, some health insurance plans will not pay the costs for people taking part in studies. Check with your health plan or insurance company to find out what they will pay for. Taking part in this study may or may not cost your insurance company more than the cost of getting regular treatment. If your insurance does not pay, you will be responsible for the charges of your regular medical care. Before you decide to participate in the study, you should check with your health insurance company to find out exactly what it will pay for.

If you have any questions about insurance coverage, including any out of pocket expenses you might incur, or which laboratory or facilities you are allowed to have tests at, a financial counselor will be made available to you upon request.

#### Will you be paid to take part in this study?

You will not receive any payment for your participation in this study.

#### How will information about you be kept private or confidential?

All efforts will be made to keep your personal information in your research record confidential, but total confidentiality cannot be guaranteed. Your personal information may be given out if required by law.

Information about your cancer and treatment will be collected from your medical record for the study. The information will be with a study identification number and stored in a secured electronic file. The electronic file is password protected and accessible only to authorized study personnel.

If information from this study is published or presented at scientific meetings, your name and

other personal information will not be used.

A description of this clinical trial will be available on <u>ClinicalTrials.gov</u>, as required by U.S. law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

# What will happen if you are injured during this study?

Subjects in this study will be exposed to certain risks of personal injury in addition to those associated with standard forms of treatment, which were discussed in the Risk and Discomforts section of this consent form. In addition, it is possible that during the course of this study, new adverse effects of paclitaxel, carboplatin, pembrolizumab and radiation therapy that result in personal injury may be discovered. The University will make appropriate referrals for medical and/or dental treatment for subjects who sustain personal injuries or illnesses as a direct consequence of participation in the research. The subject's health insurance carrier or other third-party payer will be billed for the cost of this treatment; provided that the University shall not submit to federally funded programs, e.g., Medicare, Medicaid or CHAMPUS, for reimbursement first if submission to such programs is prohibited by law. No financial compensation will be provided by the University and no other type of assistance is available from the University.

You are not giving up any of your legal rights by signing this informed consent form or by taking part in this research study.

# What will happen if you do not wish to take part in the study or if you later decide not to stay in the study?

You can decide to stop at any time. If you decide to stop for any reason, you must let the study doctor know as soon as possible so you can stop safely.

If you do not want to enter the study or decide to stop participating, your relationship with the study staff will not change, and you may do so without penalty and without loss of benefits to which you are otherwise entitled.

It is important to tell the study doctor if you are thinking about stopping so any risks from the study can be evaluated by your doctor. Another reason to tell your study doctor that you are thinking about stopping is to discuss what follow-up care and testing could be most helpful for you.

In addition, the study doctor may stop you from taking part in this study at any time if he/she believes it is in your best interest; if you do not follow the study rules; or if the study is stopped.

If you stop, you can decide whether or not to let the study doctor continue to provide your medical information to the organization running the study, however, the FDA requires that any information collected up to the point of your withdrawal cannot be removed from the study.

You may also withdraw your consent for the use of data already collected about you, but you must do this in writing to:



8

At any time, the study doctor can take you out of this study because it would not be in your best interest to stay in it, even if you are willing to stay in the study.

If you decide to withdraw from the study for any reason, you may be asked to return for at least one additional visit for safety reasons.

#### Who can you call if you have any questions?

If you have any questions about taking part in this study or if you feel you may have suffered a research related injury, you can call the study doctor:



Telephone: (732) 235-8675

If you have any questions about your rights as a research subject, you can call: IRB Director

### What are your rights if you decide to take part in this research study?

You have the right to ask questions about any part of the study at any time. You should not sign this form unless you have had a chance to ask questions and have been given answers to all of your questions.

# PERMISSION (Authorization) TO USE OR SHARE HEALTH INFORMATION THAT IDENTIFIES YOU FOR A RESEARCH STUDY

Information about you and your health is personal and private, so this information generally cannot be used in research without your written permission. The next few paragraphs tell you about how researchers want to use and share your health information in this research study. Your information will only be used as described here or as allowed or required by law. Ask questions if you do not understand any part of the research or the use of your health information. If you sign this consent form, you agree to let the researchers use your information in the research and share it with others as described below.

#### What is the purpose of the research and how will my information be used?

You are being invited to take part in this research study which is described at the beginning of this form. The purpose of collecting and using your health information for this study is to help researchers answer the questions that are being asked in the research.

#### What information about me will be used?

If you choose to be in this study, the study doctor will get your personal and medical information. This information may include:

- All information in a medical record
- Results of physical examinations
- Medical history
- Current and past medications or therapies

PI:

- Lab tests, or certain health information indicating or relating to a particular condition as well diaries and questionnaires
- · Records about study medication or drugs
- Records of blood tests
- Results of chest x-ray
- Results of imaging studies, including: MRI, CT and X-ray scans
- Information about any side effects you may experience while on study

### Who may use, share or receive my information?

The research team may use or share your information collected or created for this study with the following people and institutions:

- The \_\_\_\_\_\_ Institutional Review Board (IRB), a group of people who review the research study to protect your rights
- Officials of the
- Members of the research team, including the study doctors, research nurses and study coordinators
- the company that supplies pembrolizumab for use in this study
- The U.S. Food and Drug Administration (FDA)
- Department of Health and Human Services (DHHS) agencies
- Office of Human Research Protections (OHRP), involved in keeping research safe for people;
- Governmental agencies in other countries

Those persons or organizations that receive your information may not be required by Federal privacy laws to protect it and may share your information with others without your permission, if permitted by the laws governing them.

# Will I be able to review my research record while the research is ongoing?

No. We are not able to share information in the research records with you until the study is over. To ask for this information, please contact the Principal Investigator, the person in charge of this research study.

## Do I have to give my permission?

No. You do not have to permit use of your information. But, if you do not give permission, you cannot take part in this research study. (Saying no does not stop you from getting medical care or other benefits you are eligible for outside of this study.)

If I say yes now, can I change my mind and take away my permission later?

Yes. You may change your mind and not allow the continued use of your information (and to stop taking part in the study) at any time. If you take away permission, your information will no longer be used or shared in the study, but we will not be able to take back information that has already been used or shared with others. If you say yes now but change your mind later for use of your information in the research, you must write to the researcher and tell him of your decision:



Title: Moving PD-1 Blockade with Pembrolizumab into Concurrent Chemoradiation for Locally Advanced Non-Small Cell Lung Cancer

How long will my permission last?

There is no set date when your permission will end. Your health information may be studies for many years.

Where can you get more information?

You may call the National Cancer Institute's Cancer Information Service at: Voice: 1-800-4-CANCER (1-800-422-6237)

You may also visit the NCI Web site at http://cancer.gov/

For NCI's clinical trials information, go to: <a href="http://cancer.gov/clinicaltrials/">http://cancer.gov/clinicaltrials/</a>

For NCI's general information about cancer, go to http://cancer.gov/cancerinfo/

If you do not have access to a personal computer, you may access these websites and other information at a computer in the Resource and Learning Center on the second floor of the at no cost to you.

#### AGREEMENT TO PARTICIPATE

I agree to take part in this study.

I have read this entire form, or it has been read to me, and I believe that I understand what has been discussed. All of my questions about this form or this study have been answered.

| Subject Name: | |
|---|---|
| Subject Signature: | Date: |
| FOR NON-ENGLISH SPEAKING SUBJECTS: | |
| Signature of Reader/Translator If the Subject D | oes Not Read English Well: |
| The person who has signed above,well. You read English well and are fluent inlanguage), a language that the subject (his/her par understand the content of this consent form and parent(s)/legal guardian) the entire content of this for (his/her parent(s)/legal guardian) understands the c to ask questions regarding the consent form and the (his/her parent(s)/legal guardian). | rent(s)/legal guardian) understands well. You you have translated for the subject (his/herorm. To the best of your knowledge, the subject ontent of this form and has had an opportunity |
| Reader/Translator Name: | |
| Reader/Translator Signature: | Date: |
| Witness Name: | |
| Witness Signature: | Date: |

| Title: Moving PD-1 Blockade with Pembrolizumab into Concurrent Chemoradiation for Locally Advanced Non-<br>Small Cell Lung Cancer |
|---|
| Signature of Investigator/Individual Obtaining Consent: To the best of your ability, you have explained and discussed the full contents of the study including all of the information contained in this consent form. All questions of the research subject and those of his/her parent or legal guardian have been accurately answered. |
| Investigator/Person Obtaining Consent: |
| Signature:Date: |